CLINICAL TRIAL: NCT00061425
Title: Phase I/II Radioimmunotherapy of Non-Hodgkin's Lymphoma With Radiolabeled Humanized Immuno-LL2: Treatment With 90Y-hLL2 IgG
Brief Title: Treatment of Non-Hodgkin's Lymphoma With 90Y-hLL2 IgG
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM-T-hLL2-06-EU
Record Dates: First submitted 2003-05-27; First posted 2003-05-28 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2009-01

CONDITIONS: Non-Hodgkin's Lymphoma; Lymphoma, B-Cell
Keywords: NHL; recurrent B-cell lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: radiolabeled epratuzumab

SUMMARY:
The purpose of this trial is to determine the safety of a 90Y-radiolabeled, humanized (CDR-grafted) form of the LL2 monoclonal antibody in patients with Non-Hodgkin's lymphoma (NHL) at different dose levels.

ELIGIBILITY:
Inclusion:

* Histological or cytological diagnosis of B-cell lymphoma, and has failed at least one regimen of standard chemotherapy. (All histological grades of NHL will be eligible for this trial.)
* Measureable via CT, with at least one lesion > or = 1.5cm in one or both dimensions. (Splenic tumors in absence of other tumors will not qualify.)
* Radiological studies (ie - CT) must be performed within 4 weeks prior to study start.
* Acceptable tumor burden that will allow adequate follow-up and evaluation.
* Less that 25% bone marrow involvement, determined by bone marrow biopsy.
* Must observe the following washout periods:

At least 4 weeks beyond any major surgery. At least 4 weeks beyond any radiation therapy to the index lesion, and has recovered from radiation-induced toxicity.

At least 4 weeks beyond chemotherapy and/or immunotherapy. At least 2 weeks beyond corticosteriod(s) use and blood counts are with laboratory criteria.

* Must have Karnofsky score >70% (or equivalent, ECOG 0-2) with expected survival of at least 6 months.
* Serum creatinine < or = 1.5mg/dl or creatinine clearance > or = 50ml/min.
* Serum bilirubin < or = 2mg/dl.
* Hemoglobin > or = 10 g/dl; WBC > or = 3000/mm3; granulocyte count > or = 150/mm3; platelet count > or = 100,000/mm3 with out transfusions or cytokines for at least 30 days prior to study.
* Immunomedics ELISA assay of HahLL2 < 100ng/ml for those with prior history of monoclonal antibody infusions.
* Cognizant informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Wegener, Study Director — Gilead Sciences